CLINICAL TRIAL: NCT00035178
Title: Pharmacokinetics and Pharmacodynamics of Argatroban Injection in End-Stage Renal Disease (ESRD) Patients Undergoing Hemodialysis
Brief Title: Pharmacokinetics/Pharmacodynamics of Argatroban Injection in End-Stage Renal Disease Patients Undergoing Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Biotechnology Corporation (Industry)
Organization: Encysive Pharmaceuticals (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ARG-402
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Kidney Failure, Chronic; Renal Disease, End-Stage
Keywords: ESRD; End-stage renal disease; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — argatroban

INTERVENTIONS:
Drug: Argatroban

SUMMARY:
The primary goals of this investigation are to provide guidance on how to dose Argatroban in patients undergoing hemodialysis and to assess the safety and tolerability of Argatroban in hemodialysis patients. The secondary goal of the study will be to assess the adequacy of anticoagulation during hemodialysis.

ELIGIBILITY:
Basic Inclusion Criteria:

1. Patients, adult men or women who are between 21 and 75 years of age who are on maintenance hemodialysis regimen for at least three (3) months prior to the study start.
2. Patients who can tolerate a hemodialysis session lasting up to 9 hours.
3. Patients who can tolerate a hemodialysis treatment with blood flow rates of 300 ml per minute.
4. Female volunteers who are not documented to be surgically sterile must be willing to abstain from sexual intercourse during the study or be willing to use intrauterine devices or 2 forms of barrier contraception for at least 7 days prior to the initial dose of study medication and continuing through the completion of the study.

Basic Exclusion Criteria:

1. Any clinically relevant abnormality identified per the investigator on the screening medical assessment or laboratory examination.
2. History of regular alcohol abuse.
3. Treatment with an investigational drug within 30 days.
4. History of drug allergy of clinical significance in the opinion of the investigator.
5. Currently taking warfarin or other anticoagulants.
6. Currently taking NSAIDs (with the exception of aspirin).
7. Individuals who are obese.
8. Any history of bleeding disorder.
9. Any subject with a screening resting systolic blood pressure >180 mmHg and/or resting diastolic blood pressure of >100 mmHg unless, in the opinion of the principal investigator, the blood pressures would not endanger the subject while participating in this trial.
10. Concurrent uncontrolled cardiovascular, hematologic, respiratory, CNS, gastrointestinal disease or chronic alcoholism.
11. Anemia defined as a hematocrit of < 30 and hemoglobin < 10g/dL.
12. Concurrently taking (within the past 30 days) phenytoin, cimetidine, rifampin, cyclosporin or tacrolimus.
13. Known hypersensitivity to Argatroban or related compounds.
14. Significant hepatic insufficiency as defined by total bilirubin greater than 1.5 mg/dL or transaminase (ALT, AST) elevations greater than 2 times the upper limit of the laboratory reference range.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2002-05; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Chicago, Section of Nephrology, Chicago, Illinois
  - DaVita Clinical Research, Minneapolis, Minnesota